CLINICAL TRIAL: NCT06178146
Title: A Prospective, Open, Randomized Controlled Stage II Trial Investigating the Efficacy and Safety of Thymosin Alpha-1 in Treating Moderate to Severe Immune-related Adverse Events
Brief Title: Thymosin Alpha-1 for irAE Secondary to ICIs
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jun Wang (Other)
Responsible Party: Sponsor-Investigator, Jun Wang, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZAD-irAE
Record Dates: First submitted 2023-12-03; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: IrAE
Keywords: immune-related adverse event; thymosin alpha 1
MeSH Terms: interventions — Thymalfasin; Immunosuppressive Agents; Prednisone; Cortisone; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tα-1 group (Experimental): Subcutaneous injection with 1.6mg Thymosin alpha 1 in combination with the conventional therapy
  Interventions: Drug: Thymosin Alpha1; Drug: Immunosuppressant
- Control group (Active Comparator): Conventional therapy includes corticosteroids and other immunosuppressants according to CSCO guidelines.
  Interventions: Drug: Immunosuppressant

INTERVENTIONS:
Drug: Thymosin Alpha1 — Based on the conventional treatment, subcutaneous injection of Tα-1 (1.6 mg, qd) in Week 1; and in Week 2, subcutaneous injection of thymalfasin 1.6 mg, 3 times a week, followed by twice a week for 1 month since Week 3.
  Other Names: thymalfasin
  Arms: Tα-1 group
Drug: Immunosuppressant — Grade 2 irAEs: corticosteroid alone Grade 3 and above irAEs: corticosteroids combined with other immunosuppressants Steroid-refractory irAE: After 48-72 hours of systemic steroid therapy, the symptoms do not improve or worsen, and the second-line immunosuppressant therapy is adopted.
  Other Names: Prednisone; Cortisone; Mycophenolate Mofetil; Tacrolimus

SUMMARY:
Thymosin alpha-1 (Tα-1) has shown clinical benefits in patients whose immune functions are severely compromised or ineffective. Therefore, this study is attempted to explore whether Tα-1 could be used as a therapeutic option for the treatment of immune-related adverse events (irAEs).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are males or females, aged 18 to 75 years;
2. Subjects who are willing to sign the informed consent forms and receive follow-up visits;
3. Subjects who are cytologically or histologically diagnosed with malignant solid tumors, including but not limited to genitourinary, gynecological, lung, liver, gastrointestinal tumors and melanoma;
4. Subjects with malignant solid tumors who have developed irAEs within 6 months of immune checkpoint inhibitor therapy (CTLA-4, PD-1 and/or PD-L1). The immune checkpoint inhibitors can be used alone, or combined with chemotherapy drugs or other ICIs;
5. Subjects with Grade 2 to 4 skin toxicity, enteritis, pneumonia and hepatitis secondary to ICIs according to CTCAE V5.0 and CSCO guidelines
6. Subjects with sufficient bone marrow functions and meet the following requirements:

(1) Hemoglobin level ≥ 90 g/L (2) Neutrophil count ≥ 1.0×10^9/L (3) Lymphocyte count ≥ 0.5×10^9/L (4) Platelet count ≥75×10^9/L (5) PT, PTT, INR≤1.5 times ULN 7. Subjects with sufficient liver functions: Child-Pugh A and B; 8. Subjects with sufficient renal function: the estimated clearance rate calculated by the Cockroft-Gault formula is ≥40mL/min; 9. Suitable pregnant women who need to take effective contraceptive measures;

Exclusion Criteria:

1. Subjects who have ever immune-related adverse events due to ICI treatment;
2. Subjects who are diagnosed with immunodeficiency disease or are receiving systemic immunosuppressive therapy;
3. Subjects who have skin damage, liver damage, lung damage, etc. caused by the progression of malignant tumors;
4. Subjects who have the thromboembolic disease, biliary tract compression, perfusion injury, opportunistic infection, and liver injury caused by non-ICI drug reactions;
5. Subjects who have abnormal laboratory indicators caused by hepatotropic viruses (such as HAV, HBC, HCV) and non-hepatotropic viruses (such as Epstein-Barr virus, cytomegalovirus, and herpes simplex virus);
6. Subjects who are diagnosed with infectious colitis (e.g., caused by infections such as bacteria, Clostridium difficile, virus, fungus, parasite, etc.);
7. Subjects who suffer from autoimmune diseases, including but not limited to autoimmune hepatitis, primary cholangitis, primary sclerosing cholangitis, rheumatoid arthritis, vitiligo, psoriasis, Crohn's disease, type I diabetes, Grave's disease, etc.;
8. Subjects who suffer from other respiratory diseases with clear etiology, including malignant pulmonary infiltration, active infection, alternative systemic pulmonary toxicity or radiation pneumonitis;
9. Subjects with any other infectious diseases of grade 3 and above;
10. Subjects who have received and used thymosin products or other immunomodulators before enrollment;
11. Subjects who are allergic to thymosin products;
12. Pregnant or breastfeeding women;
13. Subjects who have any known bacterial, fungal or viral infections that may affect their safety or study compliance as deemed by the Investigator within 2 weeks before enrollment;
14. Subjects who have any health conditions that may prevent them from participating in and complying with the procedures related to the study as deemed by the Investigator, including additional laboratory abnormalities or mental illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Symptoms relieving rate | within one week after the first injection of thymalfasin.
  The proportion of immune-related adverse events reduced by at least 1 grade within 1 week after the first injection of thymalfasin.

SECONDARY OUTCOMES:
≤G1 rate | up to 8 weeks
  The proportion of total immune-related adverse events reduced to ≤ Grade 1 within 2, 4, 6 and 8 weeks after the first injection of thymalfasin;
Median relieving time | 8 weeks
  The median time for an immune-related adverse event reduced to ≤ Grade 1
The total dose of corticosteroid | 8 weeks
  The total dose of corticosteroids used during treatment, the duration and the proportion of intravenous infusion (IV)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, Professor, Principal Investigator — Shandong First Medical University
Locations (1):
- The first affiliated hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Serafino A, Pierimarchi P, Pica F, Andreola F, Gaziano R, Moroni N, Zonfrillo M, Sinibaldi-Vallebona P, Garaci E. Thymosin alpha1 as a stimulatory agent of innate cell-mediated immune response. Ann N Y Acad Sci. 2012 Oct;1270:13-20. doi: 10.1111/j.1749-6632.2012.06707.x. PMID 23050812
- [Result] Romani L, Oikonomou V, Moretti S, Iannitti RG, D'Adamo MC, Villella VR, Pariano M, Sforna L, Borghi M, Bellet MM, Fallarino F, Pallotta MT, Servillo G, Ferrari E, Puccetti P, Kroemer G, Pessia M, Maiuri L, Goldstein AL, Garaci E. Thymosin alpha1 represents a potential potent single-molecule-based therapy for cystic fibrosis. Nat Med. 2017 May;23(5):590-600. doi: 10.1038/nm.4305. Epub 2017 Apr 10. PMID 28394330
- [Result] Renga G, Bellet MM, Pariano M, Gargaro M, Stincardini C, D'Onofrio F, Mosci P, Brancorsini S, Bartoli A, Goldstein AL, Garaci E, Romani L, Costantini C. Thymosin alpha1 protects from CTLA-4 intestinal immunopathology. Life Sci Alliance. 2020 Aug 14;3(10):e202000662. doi: 10.26508/lsa.202000662. Print 2020 Oct. PMID 32817121
- [Result] Wu J, Zhou L, Liu J, Ma G, Kou Q, He Z, Chen J, Ou-Yang B, Chen M, Li Y, Wu X, Gu B, Chen L, Zou Z, Qiang X, Chen Y, Lin A, Zhang G, Guan X. The efficacy of thymosin alpha 1 for severe sepsis (ETASS): a multicenter, single-blind, randomized and controlled trial. Crit Care. 2013 Jan 17;17(1):R8. doi: 10.1186/cc11932. PMID 23327199
- [Result] Liu J, Shen Y, Wen Z, Xu Q, Wu Z, Feng H, Li Z, Dong X, Huang S, Guo J, Zhang L, Chen Y, Li W, Zhu W, Du H, Liu Y, Wang T, Chen L, Teboul JL, Annane D, Chen D. Efficacy of Thymosin Alpha 1 in the Treatment of COVID-19: A Multicenter Cohort Study. Front Immunol. 2021 Aug 2;12:673693. doi: 10.3389/fimmu.2021.673693. eCollection 2021. PMID 34408744
- [Result] Liu F, Qiu B, Xi Y, Luo Y, Luo Q, Wu Y, Chen N, Zhou R, Guo J, Wu Q, Xiong M, Liu H. Efficacy of Thymosin alpha1 in Management of Radiation Pneumonitis in Patients With Locally Advanced Non-Small Cell Lung Cancer Treated With Concurrent Chemoradiotherapy: A Phase 2 Clinical Trial (GASTO-1043). Int J Radiat Oncol Biol Phys. 2022 Nov 1;114(3):433-443. doi: 10.1016/j.ijrobp.2022.07.009. Epub 2022 Jul 21. PMID 35870709